CLINICAL TRIAL: NCT03109691
Title: Dexamethasone Effect Using Ultrasound Guided Bilateral Superficial Cervical Block for Postoperative Pain Therapy in Thyroid Surgery
Brief Title: Ultrasound Guided Bilateral Superficial Cervical Block for Post-operative Pain Therapy in Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01003060468
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-06

CONDITIONS: Bilateral Superficial Cervical Block
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): 30 patients will receive bupivacaine
  Interventions: Drug: bupivacaine; Drug: Dexamethasone; Device: ultrasound
- group 2 (Active Comparator): 30 patients will receive bupivacaine and Dexamethasone. .
  Interventions: Drug: bupivacaine; Device: ultrasound

INTERVENTIONS:
Drug: bupivacaine — group 1
Drug: Dexamethasone — group 2
  Arms: group 1
Device: ultrasound — in all groups

SUMMARY:
Ultrasound Guided Bilateral Superficial Cervical Block for Postoperative Pain Therapy in Thyroid Surgery

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I and II

Exclusion Criteria:

* allergy to local anesthetics, bleeding diatheses, and local infection or sepsis thyrotoxicosis and , malignancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | through first 24 h postoperative.
  visual analoge scale (VAS)

SECONDARY OUTCOMES:
HEART RATE | 5,10,15,30,60,90,120 min introperative
  heart rate( beats per minute)
postoperative nausea, vomiting | through first 24h postoperative
  postoperative nausea, vomiting was recorded
The time period for the first analgesic requirement | through first 24h postoperative
  total dose
blood pressure | 5,10,15,30,60,90,120 min intraoperative
  blood pressure (mm Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt